CLINICAL TRIAL: NCT05973032
Title: Minimal Residual Disease Detection by Next-generation Sequencing of Different Immunoglobulin Gene Rearrangements in Pediatric B-ALL
Brief Title: MRD Detection by NGS in Pediatric B-ALL
Status: Completed | Type: Observational
Sponsor: The Children's Hospital of Zhejiang University School of Medicine (Other)
Responsible Party: Principal Investigator, Xiaojun Xu, Principal investigator, The Children's Hospital of Zhejiang University School of Medicine
Other Study IDs: 2023-IRB-0062
Record Dates: First submitted 2023-07-25; First posted 2023-08-02 (Actual); Last update posted 2024-01-24 (Actual); Status verified 2023-07

CONDITIONS: Acute Lymphoblastic Leukemia, Pediatric
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- MRD positive and MRD negative groups: MRD postive: NGS-MRD>=0.01% at the end of induction or >=0.0001% at the end of consoidation.
  MRD negative: NGS-MRD<0.01% at the end of induction or <0.0001% at the end of consoidation.
  Interventions: Other: MRD

INTERVENTIONS:
Other: MRD — Calculate the 3-year EFS based on the MRD status (MRD positive and negative groups)

SUMMARY:
This retrospective analysis aims to investigate pediatric patients with B-cell acute lymphoblastic leukemia who were detected for minimal residual disease (MRD) using next-generation sequencing (NGS). The study will utilize second-generation sequencing technology to analyze the rearrangement of the immunoglobulin heavy chain (IGH), immunoglobulin kappa light chain (IGK), and immunoglobulin lambda light chain (IGL) genes in these patients. Patients will be stratified based on NGS-MRD levels, and the relationship between NGS-MRD and Event-Free Survival (EFS) will be evaluated.

DETAILED DESCRIPTION:
Study Design, Patients, and Procedures This was a prospective, single-center, observational study conducted in children with ALL between November 2018 and June 2022. Children with newly diagnosed B-ALL who undergone NGS of B-cell receptors at the Children's Hospital of Zhejiang University School of Medicine were included in this study.

The European Group for the Immunological Characterization of Leukemias (EGIL) criteria were applied to diagnose and classify ALL in this study. All enrolled patients were treated according to the ZJCH-ALL-2019 protocol detailed in the supplementary file. This protocol was implemented in our center in September 2018 and subsequently extended to all of Zhejiang Province in 2019. In this protocol, NGS-MRD was not used for patient risk stratification or treatment allocation. For the detection of MRD, bone marrow (BM) aspiration for Ig NGS was collected at diagnosis, the end of induction (EOI) at the 5th week from the initial prednisone prephase, and the end of consolidation (EOC) at the 13th week which was before the start of early intensification for low and intermediate risk patients, and was before the start of the second course of consolidation for high-risk patients. NGS-MRD was sequentially monitored every 2 to 3 months after consolidation until it was undetectable. In this study, NGS-MRD refers to the quantitative value of MRD detected through NGS testing which was the sum of IGH and light chain (IGK/IGL) levels. NGS detection during other timepoints, such as the interim of induction and timepoints after NGS-MRD was negative, was not mandatory but monitored as per parents' preference. The patients were followed up until August 30, 2022 and the median follow-up time was 20.7 months.

Statistical Analysis The association between categorical variables was tested using χ2 test, the correlation between quantitative variables was measured using Pearson correlation and tested using Student's t distribution, and ANOVA was used to compare quantitative variables. Event-free survival (EFS) and overall survival (OS) curves were estimated using the Kaplan-Meier method and compared according to the log rank test. Death during induction, abandonment before complete remission, death in continuous complete remission, relapse, and secondary malignancies were considered as events in the calculation of EFS probability. The EFS time was calculated from the date of diagnosis to the last date of follow-up or the first event. The OS was calculated from the date of diagnosis to death from any causes with censoring the patients alive at the time of data analysis. The final date for follow-up was August 30, 2022. Data visualization was performed using R package ggplot2 (Version 4.0.3) and GraphPad Prism 9.0.0. Statistical analysis was performed on R (Version 4.0.3). A P value of <0.05 (2 tailed) was considered to be statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* Children with newly diagnosed B-ALL who undergone NGS of B-cell receptors
* Children older than 1 year receive treatment according to the ZJCH-ALL-2019 protocol, while children younger than 1 year receive treatment according to the infant leukemia protocol.

Exclusion Criteria:

* B-cell acute lymphoblastic leukemia (B-ALL) patients who have not undergone high-throughput sequencing.
* Treated according to other protocols.

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children under the age of 18 years diagnosed with acute B-cell lymphoblastic leukemia between 2018 and 2022.
Sampling Method: Probability Sample
Enrollment: 430 (Actual)
Dates: Start 2018-11-01 (Actual); Primary Completion 2022-08-31 (Actual); Study Completion 2022-08-31 (Actual)

PRIMARY OUTCOMES:
event-free survival | Between November 2018 and June 2022
  The EFS time was calculated from the date of diagnosis to the last date of follow-up or the first event.

CONTACTS AND LOCATIONS:
Locations (1):
- The Children's Hospital of Zhejiang University School of Medicine, Hangzhou, Zhejiang, China